CLINICAL TRIAL: NCT04325490
Title: A Randomized Controlled Trial of Efficiency and Safety of Liquid Powder Containing Tapioca Starch Stimutex AS, Aloe Barbadensis, Rose Hip Oil and Allantoin Comparing With Topical 1% Hydrocortisone Cream for Treatment of Intertrigo
Brief Title: Tapioca Starch Stimutex AS, Aloe Barbadensis, Rose Hip Oil, Allantoin Comparing With Topical 1% Hydrocortisone Cream
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: HOE pharmaceuticals Sdn. Bhd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ezerra intertrigo
Record Dates: First submitted 2020-02-02; First posted 2020-03-27 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Intertrigo
Keywords: Intertrigo; Tapioca starch; Stimutex AS; Aloe barbadensis; Rose hip oil; Allantoin
MeSH Terms: conditions — Intertrigo | interventions — FR dental filling

STUDY DESIGN:
Intervention Model Description: A double-blined, randomized study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the two interventions were prepared in an identical neutral package. The same investigator evaluated the skin condition at each follow-up visit. Patients were followed up at 2 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid powder (Experimental): Liquid powder containing tapioca starch stimutex AS, aloe barbadensis, rose hip oil and allantoin on the selected intertrigo area.
  Interventions: Drug: Liquid powder
- Hydrocortisone (Active Comparator): 1% hydrocortisone cream
  Interventions: Drug: Hydrocortisone cream 1%

INTERVENTIONS:
Drug: Liquid powder — apply the study drug 1 fingertip unit to cover intertrigo lesion twice a day for two weeks.
  Arms: Liquid powder
Drug: Hydrocortisone cream 1% — apply the study drug 1 fingertip unit to cover intertrigo lesion twice a day for two weeks.
  Arms: Hydrocortisone

SUMMARY:
A randomized controlled trial of efficiency and safety of liquid powder containing tapioca starch stimutex AS, aloe barbadensis, rose hip oil and allantoin comparing with topical 1% hydrocortisone cream for the treatment of intertrigo

DETAILED DESCRIPTION:
Intertrigo is an inflammatory dermatosis involving body folds that develops through friction of skin to skin and is influenced by moist conditions. The prevalence of intertrigo was reported to be 2.5% for adults with an average age of 41.5 years. Prevalence of intertrigo in the large skin folds varies from 6% in hospital patients to 17% in nursing home clients and 20% in home care patients. The inframammary fold was most often affected (9.9%), followed by the inguinal region (9.4%), axilla (0.5%) and abdominal region (0.5%). Intertrigo may be mild and asymptomatic, but also may lead to intense erythema and desquamation. The affected skin may have a foul odor and may be macerated and ulcerated with copious or purulent discharge. The conventional therapy for simple intertrigo is minimizing moisture and friction. Some suggest the use of absorptive powders, such as talc and cornstarch, or barrier creams. These topical treatments such as topical steroid, however, have little or no proven benefit and may cause irritation or facilitate yeast colonization. This study aims to evaluate the efficacy and safety of liquid powder containing tapioca starch stimutex AS, aloe barbadensis, rose hip oil and allantoin comparing with topical 1% hydrocortisone cream of mild to moderate intertrigo patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had age more than 18 years
2. One intertrigo lesion at inframammary fold, inguinal region, interdigital, axilla or abdominal region with mild to moderate which only has erythema no epidermal loss
3. Being diagnosed intertrigo by dermatologist. Patients will be clinical and investigational with KOH preparation and Wood's lamp diagnosed with intertrigo by dermatologist.

Exclusion Criteria:

1. Patients receive topical steroids, topical anti-fungal drugs within 2 weeks prior the study
2. Patients with skin conditions including fungal/bacterial infection, Hailey-Hailey disease, pemphigus, granuloma, psoriasis, acanthosis, or Darier disease on intertriginous areas within 2 weeks prior to the study
3. Patients with an allergic to tapioca starch และ stimutex AS, aloe Barbadensis, rosa hip oil และ allantoin, or topical hydrocortisone
4. Pregnant or breastfeeding women
5. Patients with severe intertrigo treated with high potent topical steroid or systemic corticosteroid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of liquid powder containing tapioca starch stimutex AS, aloe barbadensis, rose hip oil and allantoin, compared to topical 1% hydrocortisone cream for the treatment of intertrigo. | 2 weeks
  Efficacy was evaluated by the number of patients with improvement in erythema scores on intertrigo lesion after treatment which were assessed by the patients and the same investigator. Erythema scores were recorded using a 4-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe) on intertrigo lesion at baseline and week 2.

SECONDARY OUTCOMES:
Side effects of liquid powder containing tapioca starch stimutex AS, aloe barbadensis, rose hip oil and allantoin, compared to topical 1% hydrocortisone cream for the treatment of intertrigo. | 2 weeks
  Side effects were calculated by the percentage of patients developed any side effects such as dryness, scaling, atrophy, and telangiectasia at week 2.
Patients' satisfction of liquid powder containing tapioca starch stimutex AS, aloe barbadensis, rose hip oil and allantoin, compared to topical 1% hydrocortisone cream for the treatment of intertrigo. | 2 weeks
  Satisfaction was measured on intertrigo lesion at the end of study visit by patients using visual analog scales (VAS). The minimum score is 0 (no satisfied) and the maximum score is 10 (most satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Kanokvalai Kulthanan, M.D., Principal Investigator — Mahidol University
Locations (1):
- Department of Dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Ndiaye M, Taleb M, Diatta BA, Diop A, Diallo M, Diadie S, Seck NB, Diallo S, Ndiaye MT, Niang SO, Ly F, Kane A, Dieng MT. [Etiology of intertrigo in adults: A prospective study of 103 cases]. J Mycol Med. 2017 Mar;27(1):28-32. doi: 10.1016/j.mycmed.2016.06.001. Epub 2016 Aug 21. French. PMID 27554869
- [Background] Mistiaen P, van Halm-Walters M. Prevention and treatment of intertrigo in large skin folds of adults: a systematic review. BMC Nurs. 2010 Jul 13;9:12. doi: 10.1186/1472-6955-9-12. PMID 20626853
- [Background] Gabriel S, Hahnel E, Blume-Peytavi U, Kottner J. Prevalence and associated factors of intertrigo in aged nursing home residents: a multi-center cross-sectional prevalence study. BMC Geriatr. 2019 Apr 15;19(1):105. doi: 10.1186/s12877-019-1100-8. PMID 30987588
- [Background] Kalra MG, Higgins KE, Kinney BS. Intertrigo and secondary skin infections. Am Fam Physician. 2014 Apr 1;89(7):569-73. PMID 24695603
- [Background] Wolf R, Oumeish OY, Parish LC. Intertriginous eruption. Clin Dermatol. 2011 Mar-Apr;29(2):173-9. doi: 10.1016/j.clindermatol.2010.09.009. PMID 21396557
- [Background] Hay RJ. The management of superficial candidiasis. J Am Acad Dermatol. 1999 Jun;40(6 Pt 2):S35-42. doi: 10.1016/s0190-9622(99)70396-8. PMID 10367915
- [Background] Black JM, Gray M, Bliss DZ, Kennedy-Evans KL, Logan S, Baharestani MM, Colwell JC, Goldberg M, Ratliff CR. MASD part 2: incontinence-associated dermatitis and intertriginous dermatitis: a consensus. J Wound Ostomy Continence Nurs. 2011 Jul-Aug;38(4):359-70; quiz 371-2. doi: 10.1097/WON.0b013e31822272d9. PMID 21747256
- [Background] Janniger CK, Schwartz RA, Szepietowski JC, Reich A. Intertrigo and common secondary skin infections. Am Fam Physician. 2005 Sep 1;72(5):833-8. PMID 16156342